CLINICAL TRIAL: NCT01319201
Title: Assessment of Subclinical Atherosclerosis Using Dual-source Computed Tomography Coronary Angiography in Chinese Adults With Different Glycaemic Status
Brief Title: Subclinical Atherosclerosis Using Dual-source CT Coronary Angiography in Chinese Adults With Different Glycaemic Status
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Guang Ning/Professor, Shanghai Jiao-Tong University School of Medicine
Other Study IDs: CCEMD009
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples were collected and retained for biomarker analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Impaired glucose regulation: This group of subjects was diagnosed as impaired glucose regulation using oral glucose tolerance test.
- Type 2 diabetes: This group of subjects was diagnosed as type 2 diabetes using oral glucose tolerance test.
- Normal glucose regulation: This group of subjects was considered normal regarding glucose metabolism using oral glucose tolerance test.

SUMMARY:
Part I: Survey of Coronary Artery Calcification and Stenosis in Participants with Different Glycaemic Status

Aims:

To evaluate coronary artery calcification and stenosis in community-dwelling adults with different glycaemic status, using dual-source CT angiography (CTA)

Study Subjects and Methods:

200 adults with normal glucose regulation (NGR), 200 with impaired glucose regulation (IGR) and 200 with type 2 diabetes were recruited from an urban community of Shanghai, who then underwent a comprehensive examination including questionnaire, anthropometric measurements, biochemical analysis and CTA.

Part II: Follow-up of Cardiovascular Events and Re-evaluation of Coronary Artery Calcification and Stenosis

Aims and Methods:

To investigate the development of cardiovascular diseases in subjects recruited in part I and re-evaluate coronary artery calcification and stenosis using CTA after 3-year follow-up

To identify the predictive value of coronary artery calcification and stenosis with future risks of cardiovascular diseases and the possible development of coronary artery disorders among participants with different glycaemic status

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 70 years old
2. Gender: males and females
3. Provide written informed consent
4. Satisfactory compliance

Exclusion Criteria:

1. History of cardiovascular diseases
2. Allergy to iodine
3. Exposure to radiation within last 3 months
4. ALT more than 100IU/L, or serum creatine more than 133μmol/l [1.5mg/dl] or GFR less than 60ml/min
5. Heart rate more than 100 bpm or severe arrhythmia
6. Malignancy, myocardial infection, acute hepatitis or other major diseases

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 adults with normal glucose regulation (NGR), 200 with impaired glucose regulation (IGR) and 200 with type 2 diabetes were recruited from an urban community of Shanghai
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-04

PRIMARY OUTCOMES:
Number of participants who will develop cardiovascular events during follow-up | 3 years
  Cardiovascular events include non-fatal myocardial infarction, non-fatal stroke and cardiovascular death. The progression of coronary artery calcium and stenosis is also evaluated at the final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, M.D.; PH.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao-Tong University School of Medicine, Shanghai, China